CLINICAL TRIAL: NCT01699776
Title: Comparison of Digoxin and Ivabradine in Heart Failure With Preserved Systolic Function. Time to Rethink About Digoxin.
Brief Title: Efficacy Study of Digoxin & Ivabradine to Treat Heart Failure
Acronym: Dig&Iva
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cocco, Giuseppe, M.D. (Individual)
Collaborators: Cardiology Office, Rheinfelden, Switzerland (Other)
Responsible Party: Principal Investigator, Cocco G., M.D., M.D., FESC, Cocco, Giuseppe, M.D.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CG&PJ-Dig-Iva 2009-2012
Record Dates: First submitted 2012-09-12; First posted 2012-10-04 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2012-10

CONDITIONS: Cardiac Failure
Keywords: Digoxin; Ivabradine; with atrial fibrillation.
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine; Digoxin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Active Comparator): Ivabradine, 7,5 mg b.id. by mouth for 14-16 weeks.
  Interventions: Drug: Ivabradine
- Digoxin (Active Comparator): Digoxin 0.125 mg once a day, 5 times per week, for 12-14 weeks by mouth.
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Ivabradine — 7.5 my b.id. by mouth for 12-14 weeks
  Other Names: Procoralan
  Arms: Ivabradine
Drug: Digoxin — 1.25 mg once a day by mouth, for 12-14 weeks.
  Arms: Digoxin

SUMMARY:
It is established that at a serum concentration 0.5-0.9 ng/ml digoxin is effective in patients with heart failure, especially in the presence of atrial fibrillation (AF). It is the claimed that ivabradine by lowering heart rate reduces symptoms and improves clinical outcomes in patients with heart failure. The effect of ivabradine and digoxin in heart failure was compared.

Patients 22 patients with ischemic heart failure, AF, and diastolic dysfunction with preserved left ventricular systolic function were treated with digoxin and ivabradine for 3 months, according to a randomization cross-over design.

Collected data Medical history, physical examination, laboratory (including proBNP and serum digoxin concentrations), ECG, 6-minute walk test, and echocardiographic data (LVEF, LAVi, e/e1 ratio).

DETAILED DESCRIPTION:
Protocol This is an investigator-started study, coded GC&PJ-dig-Iva 2009-2012. The study was planned according to the Good Clinical Quality standards and the analysis was performed using an intention-to-treat method. The protocol was approved from an Ethics Committee. Selected patients gave their written informed consent. The family practitioners agreed and obtained the data and analysis. Collected data were analyzed from single-blinded investigators (without knowledge of the used test drug and time of collection).

Patients Study design: same patients were assigned to DIG or IVA for 3 months, according to a randomization cross-over design.

Tested drugs Commercial brands of digoxin and ivabradine were used. Digoxin was given by mouth at a dose of 0.125 mg/day, 5 times per week, for 3 months.

Ivabradine was given by mouth at a dose of 7.5 mg bid for 3 months.

Inclusion criteria Chronic and stable coronary artery disease Permanent atrial fibrillation. Diastolic dysfunction with maintained systolic function.

Exclusion criteria Unstable angina pectoris. Reduced systolic cardiac function (LVEF<52%). Normal diastolic function. Diabetes requiring insulin. Moderate or severe renal or hepatic dysfunction. Technically insufficient echocardiographic quality.

Collected data Medical history and concomitant medications. Physical examination was performed. Laboratory values (including proBNP and serum digoxin concentration). ECG. Echocardiography. 6-minute walk test.

Statistical Analyses Data are expressed as mean ± 1 SD. Absolute values and percent changes in relation to baseline measurements were analyzed. The 2 hypotheses tested were: null hypothesis: mu1-mu2=0.0, and alternative hypothesis: mu1-mu2>>0.0. Comparisons within groups were made using paired t tests or the non-parametric Wilcoxon signed-rank test, where appropriate. Between-group comparisons were performed by unpaired t tests or the non-parametric Mann-Whitney U test, respectively. Chi-square test or Kruskal-Wallis test were used to compare continuous normally or not normally distributed and qualitative variables, where appropriate. Multivariate analysis of variance was performed. A p value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

All patients had heart failure NYHA (New York Heart Association) class III. All had chronic and stable coronary artery disease which had been treated with percutaneous dilatation and stenting, and/or aortocoronary bypass. The pathology had induced a permanent AF and heart failure with left ventricular diastolic dysfunction and preserved systolic function. Preserved systolic function was defined by a LVEF (left ventricular ejection fraction) ≥52%. Left ventricular diastolic dysfunction was defined by a e/e1 ratio > 15 (septal spectral tissue-Doppler).

Exclusion Criteria:

Unstable myocardial ischemia, reduced systolic cardiac function (LVEF<52%), diabetes mellitus requiring insulin, moderate or severe renal or hepatic dysfunction, or technically insufficient echocardiography.

Ages: 60 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Comparative therapeutic effect. | 6 months
  Effects on symptoms and signs of cardiac failure.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cocco, MD, Principal Investigator — Cardiologist, senior lecturer
Locations (1):
- Cardiology office, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Result] Cocco G, Jerie P. Comparison between ivabradine and low-dose digoxin in the therapy of diastolic heart failure with preserved left ventricular systolic function. Clin Pract. 2013 Nov 4;3(2):e29. doi: 10.4081/cp.2013.e29. eCollection 2013 Aug 2. PMID 24765517